CLINICAL TRIAL: NCT04978935
Title: Improving Pulmonary Function The Effect of Care Protocol on the Outcomes of Patients With Thoracotomy
Brief Title: The Effect of Care Protocol on the Outcomes of Patients With Lung Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Mersin University (Other)
Responsible Party: Principal Investigator, Dilara Soydan, Nursing researcher, Mersin University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: MersinUniversityNursingFaculty
Record Dates: First submitted 2021-07-07; First posted 2021-07-27 (Actual); Last update posted 2021-07-27 (Actual); Status verified 2021-07

CONDITIONS: Patient Outcomes
Keywords: Thoracotomy; Care protocol; Nursing; Nursing care; Respiratory functions
MeSH Terms: interventions — CARE protocol

STUDY DESIGN:
Intervention Model Description: Prospective, parallel, two arm, randomized controlled,single blind
Who Masked: Participant
Masking Description: 80 patients by randomization will be divided into groups A and B. Group A will be determined as the study group and group B as the control group. The information showing the nurses included in the research sample is assigned to the A and B groups will be put in an opaque envelope. This envelope will be kept by the coordinator researcher (GAU). When the researcher (DS) goes to the patient for the application, after filling the "Informed Consent Form", she will open the envelope and find out which group the patient is in. The participants will be blinded. The researcher (DS), on the other hand, cannot be blinded due to the nature of the research. When the research is completed, the data will be transferred to the computer environment by a statistician who does not know the A and B groups, and the data will be analyzed by a statistician independent of the research and the findings will be reported.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): In the control group (n=40), interventions for the position, mobilization and spirometry of the patient are applied to all patients in the clinic where the study was conducted. However, these applications are not made in accordance with a certain order and protocol. Shoulder exercises are not routinely taught to patients. In the study, no additional application will be made to the control group other than the routine treatment and care practice of the clinic.
- Intervention (Experimental): Care protocol will be applied to the study group (n=40), starting from the first day spent in the intensive care unit.Care protocol consists of patient's position, mobilization, use of spirometer and shoulder exercises. The bed head of the patient will be raised 30°-45° in line with the application steps. In the study, the patient's in-bed and out-of-bed mobilization will be provided by considering the mobilization application steps, and the patient will be asked to stay out of bed for two hours on the 0 th day after surgery. The patient will be asked to stay out of bed for six hours from the first postoperative day until discharge. After the thoracotomy, the conditions that the doctor considers as complications will be recorded.The time of chest tube removal and the day of discharge will be recorded. In the study, the use of spirometry and shoulder exercises will be carried out by taking into account the implementation steps of the care protocol.
  Interventions: Other: Care protocol

INTERVENTIONS:
Other: Care protocol — Before starting the application, the investigator (DS) will fill out the Introductory Characteristics Form of all patients, the Pre-thoracotomy Pulmonary Function Test (PFT) section of the Patient Results Form. The PFT section will be re-evaluated on the 1st, 5th day and on the day of discharge after thoracotomy.
  Nursing interventions will be applied to the study group (n=40), starting from the 0th day (the first day spent in the intensive care unit) after the thoracotomy in line with the prepared care protocol application steps until discharge. Care protocol consists of patient's position, mobilization, use of spirometer and shoulder exercises.
  Arms: Intervention

SUMMARY:
This randomized controlled trial evaluates the effect of the care protocol, which consists of independent nursing interventions, which play an important role in accelerating the recovery process of the patient, such as the patient's position, mobilization, use of spirometry, and providing shoulder exercises after thoracotomy. The hypothesis of this research is; the care protocol applied to the patients after thoracotomy has an effect on the patients' pulmonary function tests (FVC, FEV1, FEV1/FVC) and on the mobilization of the patients, the development of complications, the time of chest tube removal and the discharge

DETAILED DESCRIPTION:
Methods: In the study, 80 patients were randomly assigned to the study and control groups. Nursing interventions will be applied to the patients included in the study group (n=40), starting from the 0th day (the first day spent in the intensive care unit) after the thoracotomy in line with the prepared care protocol application steps until discharge. maintenance protocol; It will consist of position of the patient, mobilization, use of spirometer and shoulder exercises. The primary outcome of the research is the effect of the maintenance protocol used in the improvement of respiratory function on respiratory function tests. The secondary outcome of the research is to determine the effect of the care protocol on mobilization, complication development status, chest tube removal and discharge time in patients. The results are obtained by recording PFT values on the 1st, 5th and discharge days before and after thoracotomy. Postoperative (0.,1.,2.,3.,4.,5.) days and discharge day; mobilization, complication development status, chest tube removal time and discharge date will be recorded on the Patient Results Form.

ELIGIBILITY:
Inclusion Criteria:

* Accepting to participate in the research,
* 18 years and older,
* Conscious, oriented and cooperative,
* Able to speak and understand Turkish,
* Does not have any psychiatric disease,
* Elective thoracotomy performed,
* Chest tube inserted,
* Patients who were followed up in the intensive care unit on the first day after surgery and admitted to the clinic the next day
* Patients without a history of metastatic disease

Exclusion Criteria:

* Those who do not accepted to participate in the research,
* Under 18 years of age,
* Unconscious, without orientation and cooperation,
* Who cannot speak or understand Turkish,
* Having a psychiatric problem,
* Non thoracotomy
* Non chest tube,
* Metastatic disease,
* Emergency thoracotomy applied,
* Patients staying in the intensive care unit for more than one day.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-08-28 (Estimated); Primary Completion 2022-08-28 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Pulmonary function test values evaluated using the care protocol | Change from before implementation preoperative and postoperative (1.,5.) days and an average of 2 weeks
  Pulmonary function tests. Pulmonary function tests will be measured with a portable pulmonary function tester. In the evaluation, FVC (%), FEV1 (%) and FEV1/FVC (%) parameters will be used

SECONDARY OUTCOMES:
Mobilization evaluated using the care protocol | Change from before implementation and postoperative (0.,1.,2.,3.,4.,5.) days and an average of 2 weeks
  In the study, the patient's in-bed and out-of-bed mobilization will be provided by considering the mobilization application steps, and the patient will be asked to stay out of bed for two hours on the 0 th day after surgery. In the clinic, the patient will be mobilized in line with the mobilization application steps. The patient will be asked to stay out of bed for six hours from the first postoperative day until discharge. The steps taken will be recorded with the pedometer
Prevention of complications evaluated using the care protocol | Change from before implementation and postoperative (0.,1.,2.,3.,4.,5.) days and an average of 2 weeks
  After the thoracotomy, the conditions that the doctor considers as complications (atelectasis, pneumonia, air leak, bronchospasm, subcutaneous emphysema, atrial fibrillation) will be recorded and daily evaluation will be made.
Chest tube removal evaluated using the care protocol | Change from before implementation and postoperative (0.,1.,2.,3.,4.,5.) days and an average of 2 weeks
  The time of chest tube removal and the day will be recorded in the Patient Results Form
Discharge time evaluated using the care protocol | Change from before implementation and postoperative (0.,1.,2.,3.,4.,5.) days and an average of 2 weeks
  The time of discharge will be recorded in the Patient Results Form

CONTACTS AND LOCATIONS:
Overall Officials: GÜLAY ALTUN UĞRAŞ, Doctorate, Study Director — Researcher

IPD SHARING:
Plan to Share IPD: No